CLINICAL TRIAL: NCT05860348
Title: Symptomatic CRT Patients: Real-World Experience - Barostim™ Advancing the Level of Clinical Evidence. A Post-Market Registry With the Barostim™ System
Brief Title: Symptomatic CRT Patients: Real-World Experience - Barostim™ Advancing the Level of Clinical Evidence
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 360064-001
Record Dates: First submitted 2023-04-18; First posted 2023-05-16 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Device: Barostim™ System: Implantation of the Barostim™ System
  Interventions: Device: Barostim™ System

INTERVENTIONS:
Device: Barostim™ System — Implantation of the Barostim™ System

SUMMARY:
The purpose of this study is to develop valid scientific evidence of the safety and benefit of Barostim Therapy in the commercial setting in patients that are symptomatic despite having received CRT.

DETAILED DESCRIPTION:
This is a non-randomized, prospective, multicenter complementary-study of the REBALANCE Registry. Patients who have been implanted with a CRT device at least 6-months prior to enrollment are eligible for this complementary-study. Up to 150 subjects will be enrolled. Data should be obtained from evaluations taken prior to implant, at implant, and every six months after device implant, up to the 36-month visit at which time each patient will be exited from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients can be included if they were implanted with a cardiac resynchronization therapy (CRT) device at least six months (180 days) prior to informed consent and are planned for a de novo Barostim System implantation. Patients must sign an informed consent form before implantation with the Barostim System in order to participate in this study.

Exclusion Criteria:

* Patients cannot be enrolled and active in another (e.g. device, pharmaceutical, or biological) clinical study unless approved by the CVRx Clinical department.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Heart failure patients who have been implanted with a CRT device and are planned for a de novo Barostim System implantation.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Change in Six Minute Hall Walk | 36 months post-implant
  Changes in Six Minute Hall Walk distance through 36 months post-implant

SECONDARY OUTCOMES:
Change in Minnesota Living with Heart Failure Quality of Life | 6 months post-implant
  Changes in Minnesota Living with Heart Failure Quality of Life through 6 months post-implant
Change NYHA Class | 6 months post-implant
  Changes in NYHA Classification through 6 months post-implant

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Florida Heart Rhythm Specialists, Fort Lauderdale, Florida
  - Advanced Cardiology, Hackettstown, New Jersey

IPD SHARING:
Plan to Share IPD: No